CLINICAL TRIAL: NCT04491981
Title: Longevity of Restoration Repairs Using Composite Resin Versus High Viscosity Glass Ionomer in Primary Molars: Randomized Clinical Trial
Brief Title: Restoration Repairs Using Composite Resin Versus Glass Ionomer in Primary Molars: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Professor Doctor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REPAIRC3
Record Dates: First submitted 2020-06-15; First posted 2020-07-30 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Dental Caries; Dental Caries in Children
MeSH Terms: conditions — Dental Caries | interventions — Composite Resins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encapsulated Glass Ionomer Cement (Experimental): Repair of restorations in primary molars using a high viscosity glass ionomer cement (RIVA Self Cure - SDI)
  Interventions: Procedure: Encapsulated Glass Ionomer Cement
- Composite resin (Experimental): Repair of restorations in primary molars using a composite resin (Filtek Bulk Fill- 3M ESPE)
  Interventions: Procedure: Composite resin

INTERVENTIONS:
Procedure: Encapsulated Glass Ionomer Cement — Repair of restorations in primary molars using Encapsulated High Viscosity Glass Ionomer (RIVA Self Cure - SDI). No local anesthesia will be used. A portion of the former restoration and infected carious tissue can be removed if necessary, and then the restoration will be repaired with GIC (Glass Ionomer Cement).
  Arms: Encapsulated Glass Ionomer Cement
Procedure: Composite resin — Repair of restorations in primary molars using composite resin (Filtek Bulk Fill- 3M ESPE.) No local anesthesia will be used.A portion of the former restoration and infected carious tissue can be removed if necessary, and then the restoration will be repaired with CR (composite resin).
  Arms: Composite resin

SUMMARY:
The objective of this randomized clinical study is to evaluate the survival of repairs in restorations using composite resin (CR) or high viscosity glass ionomer cement (GIC) in primary molars. This trial is nested to another study (NCT03520309), so patients will be enrolled from CARDEC 3. 312 restorations will be included and randomized into two groups: glass ionomer cement (Riva Self Cure, SDI, Australia) and composite resin (Filtek Bulk Fill and Filtek Bulk Fill Flow, 3M ESPE, USA). After the end of treatments, patients will be followed for 24 months to assess the success of the restorations, which will be considered as the absence of the need for reintervention. The Kaplan-Meier survival curves and the log-rank tests will be performed to assess survival between groups and Cox regression analysis will be used to compare the outcome with the variables (α = 5%).

DETAILED DESCRIPTION:
Failed restorations in primary teeth will be repaired using GIC or composite resin.

ELIGIBILITY:
Inclusion Criteria:

* Children who have sought treatment in the School of Dentistry, University of Sao Paulo
* Children between 3 and 10 years old
* Children presenting at least one restoration (of any material, any surface and any integrity status) in primary teeth

Exclusion Criteria:

* Children whose parents did not agree to participate in the study
* Children with behavioural issues at the initial exam or who did not assent to participate in the study

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success of restorations after repair | 24 months
  Visual assessment using Frencken criteria for occlusal restoration and Roeleveld et al. criteria for occlusoproximal restorations

SECONDARY OUTCOMES:
Cost- effectiveness of restorations repairs | 24 months
  To assess this outcome measure we will consider the percentage of patients needing new operatory interventions and costs will be assessed in monetary units (US dollars)
Patient's discomfort | baseline
  Wong-Baker facial scale - from 0 to 5 (immediately after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - School of Dentistry, São Paulo, Brazil

REFERENCES:
- [Background] Opdam NJ, van de Sande FH, Bronkhorst E, Cenci MS, Bottenberg P, Pallesen U, Gaengler P, Lindberg A, Huysmans MC, van Dijken JW. Longevity of posterior composite restorations: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):943-9. doi: 10.1177/0022034514544217. Epub 2014 Jul 21. PMID 25048250
- [Background] Moncada G, Vildosola P, Fernandez E, Estay J, de Oliveira Junior OB, de Andrade MF, Martin J, Mjor IA, Gordan VV. Longitudinal results of a 10-year clinical trial of repair of amalgam restorations. Oper Dent. 2015 Jan-Feb;40(1):34-43. doi: 10.2341/14-045-C. Epub 2014 Aug 6. PMID 25100406
- [Background] Gordan VV, Riley JL 3rd, Blaser PK, Mondragon E, Garvan CW, Mjor IA. Alternative treatments to replacement of defective amalgam restorations: results of a seven-year clinical study. J Am Dent Assoc. 2011 Jul;142(7):842-9. doi: 10.14219/jada.archive.2011.0274. PMID 21719808
- [Background] Fernandez E, Martin J, Vildosola P, Oliveira Junior OB, Gordan V, Mjor I, Bersezio C, Estay J, de Andrade MF, Moncada G. Can repair increase the longevity of composite resins? Results of a 10-year clinical trial. J Dent. 2015 Feb;43(2):279-86. doi: 10.1016/j.jdent.2014.05.015. Epub 2014 Jun 4. PMID 24907560
- [Background] Casagrande L, Laske M, Bronkhorst EM, Huysmans MCDNJM, Opdam NJM. Repair may increase survival of direct posterior restorations - A practice based study. J Dent. 2017 Sep;64:30-36. doi: 10.1016/j.jdent.2017.06.002. Epub 2017 Jun 8. PMID 28602850
- [Background] Kanzow P, Wiegand A, Gostemeyer G, Schwendicke F. Understanding the management and teaching of dental restoration repair: Systematic review and meta-analysis of surveys. J Dent. 2018 Feb;69:1-21. doi: 10.1016/j.jdent.2017.09.010. Epub 2017 Sep 21. PMID 28943362
- [Background] Qvist V, Poulsen A, Teglers PT, Mjor IA. The longevity of different restorations in primary teeth. Int J Paediatr Dent. 2010 Jan;20(1):1-7. doi: 10.1111/j.1365-263X.2009.01017.x. PMID 20059587
- [Background] Dias AGA, Magno MB, Delbem ACB, Cunha RF, Maia LC, Pessan JP. Clinical performance of glass ionomer cement and composite resin in Class II restorations in primary teeth: A systematic review and meta-analysis. J Dent. 2018 Jun;73:1-13. doi: 10.1016/j.jdent.2018.04.004. Epub 2018 Apr 9. PMID 29649506
- [Background] Tedesco TK, Calvo AF, Lenzi TL, Hesse D, Guglielmi CA, Camargo LB, Gimenez T, Braga MM, Raggio DP. ART is an alternative for restoring occlusoproximal cavities in primary teeth - evidence from an updated systematic review and meta-analysis. Int J Paediatr Dent. 2017 May;27(3):201-209. doi: 10.1111/ipd.12252. Epub 2016 Aug 4. PMID 27489205
- [Background] Pitts NB, Richards D. Personalized treatment planning. Monogr Oral Sci. 2009;21:128-143. doi: 10.1159/000224217. Epub 2009 Jun 3. PMID 19494680
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Ismail AI, Pitts NB, Tellez M; Authors of International Caries Classification and Management System (ICCMS); Banerjee A, Deery C, Douglas G, Eggertsson H, Ekstrand K, Ellwood R, Gomez J, Jablonski-Momeni A, Kolker J, Longbottom C, Manton D, Martignon S, McGrady M, Rechmann P, Ricketts D, Sohn W, Thompson V, Twetman S, Weyant R, Wolff M, Zandona A. The International Caries Classification and Management System (ICCMS) An Example of a Caries Management Pathway. BMC Oral Health. 2015;15 Suppl 1(Suppl 1):S9. doi: 10.1186/1472-6831-15-S1-S9. Epub 2015 Sep 15. No abstract available. PMID 26391116
- [Background] Qvist V, Poulsen A, Teglers PT, Mjor IA. Fluorides leaching from restorative materials and the effect on adjacent teeth. Int Dent J. 2010 Jun;60(3):156-60. PMID 20684440
- [Background] Gordan VV, Riley JL 3rd, Rindal DB, Qvist V, Fellows JL, Dilbone DA, Brotman SG, Gilbert GH; National Dental Practice-Based Research Network Collaborative Group. Repair or replacement of restorations: A prospective cohort study by dentists in The National Dental Practice-Based Research Network. J Am Dent Assoc. 2015 Dec;146(12):895-903. doi: 10.1016/j.adaj.2015.05.017. PMID 26610834
- [Background] Hickel R, Brushaver K, Ilie N. Repair of restorations--criteria for decision making and clinical recommendations. Dent Mater. 2013 Jan;29(1):28-50. doi: 10.1016/j.dental.2012.07.006. Epub 2012 Aug 3. PMID 22867859
- [Background] Frencken JE. Evolution of the the ART approach: highlights and achievements. J Appl Oral Sci. 2009;17 Suppl(spe):78-83. doi: 10.1590/s1678-77572009000700014. PMID 21499660
- [Background] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533
- See also: Randomization website — https://www.sealedenvelope.com/simple-randomiser/v1/